CLINICAL TRIAL: NCT05017948
Title: Alleviating Geriatric Inpatients' Medication-related Iatrogenesis
Acronym: AGING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Luigi Brunetti, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2021001087
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Iatrogenic Disease; Risk Reduction
MeSH Terms: conditions — Iatrogenic Disease; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Discharge medication regimen instructions will be provided upon discharge after being assessed using the MWRS, optimized, and assessed by the prescriber.
  Interventions: Other: Risk score based intervention
- Standard of Care (No Intervention): Discharge medication regimen instructions will be provided upon discharge after being assessed by the prescriber.

INTERVENTIONS:
Other: Risk score based intervention — Targeted interventions based off of risk score software
  Arms: Intervention

SUMMARY:
This study will evaluate the MedWise Risk Score™ (MWRS™), a holistic approach to quantifying the risk of a patient's medication regimen. High risk patients will be identified at hospital discharge. Targeted interventions will be made to reduce their MWRS™ with a 30-day follow up. The hypothesis being tested is that a reduction in MWRS™ will lead to reduced 30-day readmission.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for at least 48 hours
* Prescribed at least 5 medications at hospital discharge
* Baseline medication risk score of 20 or more

Exclusion Criteria:

* Reside greater than 25 miles from the index facility
* Discharge to hospice
* Discharge against medical advice
* Patient expiration during initial hospitalization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Number of individuals with an emergency department visit or hospital readmission | 30 days after hospital discharge
  Number of individuals with an emergency department visit or hospital readmission

SECONDARY OUTCOMES:
Difference in score between patients aged older and younger than 65 years | At time of intervention
  Comparison between age groups

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in publications, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: Data will be shared with investigators whose proposed use of the data has been approved. Proposals should be directed to brunetti@rutgers.edu.